CLINICAL TRIAL: NCT03790878
Title: Evaluating the Impact of an Emotion Regulation Intervention on Emotion Perception
Brief Title: Emotion Regulation and Emotion Perception
Acronym: EREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Mind and Life Institute, Hadley, Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00089935; 1F31MH117830-01A1 (NIH)
Record Dates: First submitted 2018-12-28; First posted 2019-01-02 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2018-12

CONDITIONS: Emotions
Keywords: Emotion Dysregulation; Empathy; Emotion Perception
MeSH Terms: interventions — Habituation, Psychophysiologic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindful Breathing (Experimental): Participants receive training in a mindful breathing skill to regulate their emotional distress during a stressor task. They will then receive one week of reminders to use this skill, delivered through their mobile phones.
  Interventions: Behavioral: Mindful Breathing
- Habituation (Active Comparator): Participants receive an exposure/habituation intervention to regulate their emotional distress during a stressor task. They will then receive one week of reminders, delivered through their mobile phones.
  Interventions: Behavioral: Habituation
- Control (Placebo Comparator): Participants complete the stressor task with no emotion regulation training. Similar to the other conditions, they will then receive one week of reminders, delivered through their mobile phones to test for placebo effects.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Mindful Breathing — Training in a mindful breathing skill that reduces emotional distress
  Arms: Mindful Breathing
Behavioral: Habituation — An exposure procedure that reduces emotional distress through habituation
  Arms: Habituation
Behavioral: Control — No emotion regulation intervention, placebo
  Arms: Control

SUMMARY:
The purpose of this study is to assess the impact of a brief, emotion regulation intervention on the ability to perceive other people's emotions.

DETAILED DESCRIPTION:
Decision to close enrollment was made on January 2, 2020.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-55;
2. have a smartphone and agree to receive text-messages;
3. have difficulty with their relationships or social interactions;
4. high emotion dysregulation, assessed with the Difficulties with Emotion Regulation Scale (DERS)(Gratz & Roemer, 2004) with scores over 90.

Exclusion Criteria:

1. Current mania;
2. Meets full criteria for any current psychotic disorder;
3. Currently/chronically homeless;
4. Current suicidal ideation;
5. Psychiatric hospitalization within past 6 months;
6. Unable to read, blind or deaf. Our previous study recruited only participants who were currently in treatment, but this study will include both participants who are currently in treatment, as well as those who are not in treatment.
7. high self-reported autistic traits, as assessed by the Autism Spectrum Quotient (Auyeung & Baron-Cohen, 2012).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Z Rosenthal, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Will check with sponsors on Duke's policies for data sharing and may update the plan in the future.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants were considered screen failures
Period: Overall Study
Arm/Group | Mindful Breathing | Habituation | Control
Started | 26 | 27 | 27
Completed | 26 | 27 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindful Breathing | Habituation | Control | Total
Number analyzed (Participants) | 26 | 27 | 27 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.56 (7.56) | 23.77 (7.03) | 23.77 (20) | 25 (6.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 20 | 64
  Male | 6 | 3 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 3 | 10
  Not Hispanic or Latino | 23 | 23 | 24 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 8 | 10 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 5 | 12
  White | 13 | 11 | 9 | 33
  More than one race | 3 | 3 | 3 | 9
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 27 | 80

OUTCOME MEASURES:

1. Primary Outcome: The Ability to Perceive Negative and Positive Emotional Expressions, as Measured by a Behavioral Computer-based Assessment
Description: Emotion perception is measured by a computer-based behavioral assessment during the laboratory session. Scores for negative emotional expressions range from 0-100%, with higher scores indicating greater emotion perception accuracy.
Time Frame: During the laboratory experiment (week 1)
Population: Baseline data for one participant was not completed appropriately and was omitted from the analysis.
Measure: Mean (Standard Deviation); unit: Percent of correct responses
Arm/Group | Mindful Breathing | Habituation | Control
Number analyzed (Participants) | 25 | 27 | 27
Percent of correct responses | 77.31 (14.36) | 81.93 (17.94) | 84.85 (16)
Statistical Analysis 1: Comparison: Mindful Breathing vs Habituation vs Control; Test type: Other; p = 0.018, ANCOVA

2. Primary Outcome: Changes in Emotion Perception, as Measured by a Phone-based Behavioral Assessment
Description: Perception of positive emotional expressions and negative emotional expressions are measured by a behavioral phone-based assessment, delivered multiple times over one week via mobile phones. Scores for ratings of emotional valence range from 0-9, with higher scores as more positive emotional valence and lower scores as more negative emotional valence.
Time Frame: After the one week of phone-based intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Breathing | Habituation | Control
Number analyzed (Participants) | 26 | 27 | 27
units on a scale | 5.19 (2.57) | 5.3 (2.54) | 5.23 (2.59)
Statistical Analysis 1: Comparison: Mindful Breathing vs Habituation vs Control; Test type: Other; p = 0.396, Multilevel modeling

3. Secondary Outcome: Change in Emotional Distress, as Measured by Subjective Units of Distress (SUDS)
Description: SUDS are measured on a 10-point Likert self-report scale of Subjective Units of Distress, ranging from 0-9. Scores are changes in SUDS ratings from before hearing the tone to after the tone, with greater scores indicating greater reductions in distress (positive outcomes). SUDS score was evaluated at the beginning of the laboratory experiment, and then at the very end of the lab experiment. The change score was calculated by subtracting the beginning score from the end score.
Time Frame: Beginning of Week one laboratory experiment, End of Week one laboratory experiment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Breathing | Habituation | Control
Number analyzed (Participants) | 26 | 27 | 27
units on a scale | 1.14 (1.21) | 0.61 (0.9) | 0.56 (0.95)
Statistical Analysis 1: Comparison: Mindful Breathing vs Habituation vs Control; Test type: Other; p = 0.002, Multilevel modeling

4. Other Pre Specified Outcome: Changes in Emotional Arousal, as Measured by Skin Conductance Response (SCR)
Description: Changes in emotional arousal are measured physiologically with electrodermal activity. Skin conductance response measures phasic changes in electrical conductivity of skin, with a minimum threshold of 0.01μS with higher values indicating greater changes in emotional arousal.
Time Frame: Laboratory assessment, up to one week
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 3 weeks. Adverse events were assessed at intake, training session, and exit.
Arm/Group | Mindful Breathing | Habituation | Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT03790878/Prot_SAP_000.pdf